CLINICAL TRIAL: NCT00583479
Title: A Prospective Study of Celiac Block Technique: One Injection or Two?
Brief Title: Prospective Study of Celiac Block Injection: 1 vs. 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Dr. Julia LeBlanc, MD, MPH, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0203-32
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Pancreatitis; Pancreatic Cancer
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): subjects who get one medication injection into the celiac ganglion during the EUS
  Interventions: Other: one injection into the celiac ganglion
- B (Other): subjects who get divided dose of the medication injected into two locations within the celiac ganglion during the EUS
  Interventions: Other: two injections into the celiac ganglion

INTERVENTIONS:
Other: one injection into the celiac ganglion — one injection into the celiac ganglion of the standard medication for CB for with chronic pancreatitis or pancreatic cancer
  Arms: A
Other: two injections into the celiac ganglion — two injection into the celiac ganglion of the standard medication for CB for with chronic pancreatitis or pancreatic cancer
  Arms: B

SUMMARY:
The purpose of this prospective randomized study is to compare the clinical effectiveness of EUS-guided CB performed with a single injection versus two injections of medication into the celiac ganglion region.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic abdominal pain from documented chronic pancreatitis or pancreatic cancer that are referred for EUS-guided celiac block will be eligible to participate in this study. Chronic pancreatitis and pancreatic cancer must be measured and documented by prior CT, ERCP, or EUS.
* Patients should not have significant co-morbidities such as uncontrolled heart failure, or severe chronic obstructive pulmonary disease (COPD) that would limit survivability of the sedation given or the procedure.
* Age > or = to 18 years
* No evidence of significant active infection (ie. pneumonia, peritonitis, wound sepsis, etc)
* No evidence of serious ongoing illness such as uncontrolled metabolic disease (diabetes mellitus, hypothyroidism, etc)
* No evidence of dementia or altered mental status that would prohibit the giving and understanding of informed consent, and no evidence of psychiatric risk that would preclude adequate compliance with this protocol.
* Patient must provide signed written informed consent.
* Patients that have had a previous celiac plexus block are eligible for this study

Exclusion Criteria:

* The patient's celiac trunk should be imaged clearly under endoscopic ultrasound. The patient's celiac plexus should be accessed easily with a needle for the medication injection. If this cannot be done safely due to the patient's anatomy (intervening blood vessel or tumor), the patient will not be eligible for the procedure or study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Compare the clinical effectiveness of EUS-guided CB performed with a single injection versus two injections of medication into the celiac ganglion region | 24-hour after the procedure; then every week thereafter until the subject is no longer in the study

SECONDARY OUTCOMES:
change in medication use | at 24-hours after procedure and every week thereafter until the subject is no longer in the study
change is pain score | at 24-hours after procedure and every week thereafter until the subject is no longer in the study
complications related to CB | at 24-hours after procedure and every week thereafter until the subject is no longer in the study

CONTACTS AND LOCATIONS:
Overall Officials: Julia LeBlanc, MD, MPH, Principal Investigator — Indiana University
Locations (1):
- Clarian Health: Indiana University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] LeBlanc JK, Al-Haddad M, McHenry L, Sherman S, Juan M, McGreevy K, Johnson C, Howard TJ, Lillemoe KD, DeWitt J. A prospective, randomized study of EUS-guided celiac plexus neurolysis for pancreatic cancer: one injection or two? Gastrointest Endosc. 2011 Dec;74(6):1300-7. doi: 10.1016/j.gie.2011.07.073. Epub 2011 Oct 13. PMID 22000795